CLINICAL TRIAL: NCT06151652
Title: Effect of Alpha-Lipoic Acid Supplementation on the Incidence of Postoperative Atrial Fibrillation in Cardiac Surgery Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ALA post cardiac surgery
Record Dates: First submitted 2023-09-24; First posted 2023-11-30 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Atrial Fibrillation
MeSH Terms: interventions — Thioctic Acid; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Control group, N = 175 patients) (Placebo Comparator): which will include patients adopted to the hospital standard of care.
  Interventions: Drug: Placebo
- Group 2 (Test group, N = 175 patients) (Active Comparator): which will include patients who will receive Alpha-lipoic acid (Thiotacid 600 mg ®) at a dose of 600 mg three times daily for one day prior to surgery, followed by Alpha-lipoic acid 600 mg twice daily for 5 days post-surgery plus the standard care.
  Interventions: Drug: Alpha Lipoic Acid 600 MG Oral Tablet

INTERVENTIONS:
Drug: Alpha Lipoic Acid 600 MG Oral Tablet — Alpha-lipoic acid (Thiotacid 600 mg ®) at a dose of 600 mg three times daily for one day prior to surgery, followed by Alpha-lipoic acid 600 mg twice daily for 5 days post-surgery plus the standard care.
  Arms: Group 2 (Test group, N = 175 patients)
Drug: Placebo — placebo
  Arms: Group 1 (Control group, N = 175 patients)

SUMMARY:
ALA is administered orally since it is without difficulty absorbed in the stomach. ALA goes through the blood brain barrier and does not show toxic effects and actions at doses used for prophylactic and therapeutic purposes. This has encouraged us to use an efficient anti-oxidant and anti-inflammatory agent, alpha-lipoic acid (biochemical) as a relevant option to prevent POAF.

DETAILED DESCRIPTION:
Investigators computed on the basis of findings from a prior study found the incidence of POAF after cardiac surgery of about 25% . Assuming a slightly lower alpha-lipoic acid' effect to previous study. If the true relative risk of AF for experimental subjects relative to controls is 0.5 , with α equivalent to 0.5 and power (1 - β) is 0.8, the estimated sample size is 152 experimental subjects and 152 control subjects in order to be able to reject the null hypothesis that this relative risk equals 1 with probability (power) of 0.8. investigators used the uncorrected chi-squared statistics to evaluate this null hypothesis. STATA software version and taking into account a possible dropout of 15%, the total sample size was: 304 + 0.15 (304) × 2 = 350 subjects of which there will be 175 controls and 175 experimental subjects %, assuming an enrolment ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* I
* Male or female patients above 18 years of age who are scheduled for cardiac surgery.

Exclusion Criteria:

* Any urgent or emergency surgery.
* Poor Left ejection volume (EF < 30%).
* Intake of steroids or any antiarrhythmic drugs except beta blockers during the last month before surgery
* Unable or unwilling to provide informed written consent.
* Pregnancy or lactation
* Known hypersensitivity to the study drug.
* Current treatment with antioxidants or alpha-lipoic acid for any indication.
* Infection or inflammatory disease except coronary artery disease.
* Left atrium size >70 mm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
• Number of Participants with POAF | 1 month

SECONDARY OUTCOMES:
Total intensive care unit length-of-stay | 3 months
  number of days at intensive care unit
Total hospital length-of-stay | 3 months
  number of days at hospital
30 days mortality | 1-month
  deaths number
Serum creatinine | 5 days
  creatinine level
Major adverse cardiovascular outcomes | 1 month
  (Myocardial injury - Stroke - Permanent pacemaker - Pericardial effusion and pleural effusion- Bleeding)
Duration of ventilation | 5 days
  hours needed to remove ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Adel, PhD, Study Director — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No